CLINICAL TRIAL: NCT05560282
Title: Fenfluramine for the Treatment of Refractory Epilepsy in Adult Dravet Patients
Brief Title: Fenfluramine for Adult Dravet Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Zogenix, Inc. (Industry)
Responsible Party: Principal Investigator, Danielle Andrade, Professor of Medicine (Neurology), Director Adult Genetic Epilepsy Program, Medical Director Epilepsy Program, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-5681
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Dravet Syndrome; Dravet Syndrome, Intractable
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fenfluramine (Experimental): Fenfluramine, oral,
  1. starting at 0.1mg/kg twice daily, maximum 26mg/day in patients not taking concomitant stiripentol
  2. starting at 0.1mg/kg twice daily, maximum 17mg/day in patients taking concomitant stiripentol
  Interventions: Drug: Fenfluramine

INTERVENTIONS:
Drug: Fenfluramine — FINTEPLA oral solution contains 2.2 mg/mL fenfluramine, equivalent to 2.5 mg/mL of the hydrochloride salt. The active ingredient, fenfluramine hydrochloride, is designated chemically as N-ethyl-α- methyl-3-(trifluoromethyl) phenethylamine hydrochloride.
  Fenfluramine hydrochloride is a white to off-white crystalline solid. The pKa of fenfluramine is 10.2. FINTEPLA is a clear, colorless solution, pH 5.
  Other Names: ZX008; Fintepla

SUMMARY:
Full Title: Fenfluramine for the treatment of refractory Epilepsy in Adult Dravet patients

Short Title: Fenfluramine for Adult Dravet patients

Clinical Phase: Phase III

Sample Size: A total of 15 participants will be included in the study.

Study Population: Adult patients (18 years and older) with drug-resistant epilepsy (maintained on their existing medications, with exception of cannabidiol) and genetically confirmed Dravet syndrome will be recruited to participate in the study.

Accrual Period: 12 months Study Design: Open label, non-randomized and uncontrolled add-on trial in adults (18 years of age and older) residing in Ontario, with refractory motor seizures and maintained on their existing antiepileptic medications, with exception of cannabidiol.

Study Duration:

• Treatment period: 12 months Study duration: 28 months

Study Agent/ Intervention/ Procedure:

Name of study drug: fenfluramine (FINTEPLA)

Dose and frequency: starting at 0.1 mg/kg twice daily, maximum 26 mg/day, in patients not taking concomitant stiripentol; starting at 0.1 mg/kg twice daily, maximum of 17 mg/day in patients taking concomitant stiripentol. All doses are divided to twice a day.

Duration:

Baseline phase: 4 weeks (no study drug) Titration phase: 2 weeks (if not taking stiripentol) to 3 weeks (if the patient is taking stiripentol) Treatment phase: 12 weeks Extension phase: up to 38 weeks, for patients who had at least a 50% decrease in seizure frequency Post-trial washout phase: 2 weeks (if not taking stiripentol) to 3 weeks (if the patient is taking stiripentol)

Route of administration:

Oral

Efficacy and safety points of interest

* Monthly convulsive seizure frequency (MCSF) reduction ≥ 50%
* Improvement in motor function
* Improvement in Cognition and Behavior
* Improvement in Quality of Sleep
* Improvement in Quality of life
* Determination of Cardiovascular safety in adults
* Responder analysis (≥25%, ≥75%, or 100% reduction in mean MCSF)
* Longest period of seizure freedom
* Number of Emergency room visits
* Use of rescue medication (number of days in 28 day-periods)
* Duration of post-ictal stage
* Frequency of other seizure types
* Body weight changes
* Patient's global functioning prior to and after study (Clinical Global Impressions Scale)

Trial registration:

www.clinicaltrials.gov

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female patients 18 years of age and older. 2. Diagnosis of DS secondary to a genetically confirmed pathogenic variant. 3. Patients recruited from the Adult Epilepsy Genetics Clinic at Toronto Western Hospital. We will also accept referrals from other academic epilepsy centers across Ontario and that are referred to our program, making this a single site study.

  4. At least 4 convulsive seizures per month at the start of the study, despite having been treated with at least two different antiepileptic drugs (given concurrently or sequentially) for at least one year.

  5. At least 4 convulsive seizures per month during the prospective Baseline Phase (4 weeks).

  6. Able to provide written consent signed by study participant's caregiver prior to entering the study or undergoing any study procedures.

  7. Participant's caregivers should be able to record seizures and report adverse events for the full duration of the study.

  8. No evidence of non-compliance with ongoing ASM therapy. 9. Stable dose(s) of the same ASMs for one month prior to screening. 10. If participant has a vagal nerve stimulator or deep brain stimulator, it must have been implanted for at least six months prior to recruitment. Stimulator parameters may not be changed for at least one month prior to screening or thereafter during the study. Magnet use will be allowed but must be documented throughout the study.

  11. Patient's caregivers agree that patient will not to take any cannabinoids or any other investigational compound for 1 month before the study or outside cannabinoids during the study.

  12. Patient's caregivers agree that patient will have blood samples taken and stored for assays.

  13. Is planning to stay in the country for the duration of the trial. 14. Can travel to the study site for the initial in-person visit with the study physicians and to a local lab for blood collection (Lifelabs).

  15. Patient's caregiver has access to telephone, computer, and internet to complete the study questionnaires.

  16. Sexually active women of child-bearing potential (WCBP) and males must be using a medically acceptable method of birth control. Women who are of non child-bearing potential, i.e., post-menopause, must have this condition captured in their medical history. A medically acceptable method of birth control includes barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge), intrauterine devices in place for at least 3 months, surgical sterilization, or adequate barrier methods (e.g., diaphragm and foam). Use of oral contraceptives in combination with another method (e.g., a spermicidal cream) is acceptable. In participants who are not sexually active, abstinence is an acceptable form of birth control.

Exclusion Criteria:

* 1. Participation in a study involving administration of an investigational compound within one month of First appointment.

  2. Evidence of clinically significant non-epileptic disease (cardiac, respiratory, gastrointestinal, hepatic, hematologic or renal disease, etc.) that in the opinion of the investigators could affect the patient's safety or trial conduct.

  3. Pulmonary hypertension (systolic pressure>35 mmHg) 4. Cardiovascular or cerebrovascular disease 5. Current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy defined as greater than moderate and/or mild aortic regurgitation on echocardiogram 6. Treatment with centrally acting anorectic agents, monoamine oxidase inhibitors or other centrally acting agent with serotonin antagonist or agonist properties.

  7. Current or past history of glaucoma 8. Hypersensitivity to FEN or any of the excipients in the study medication 9. Use of CBD oil 10. Pregnant and/or breastfeeding women are excluded from this study. Sexually active women must have negative pregnancy urine test in first in-person visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Seizure reduction | 16 week
  Comparing the proportion of participants with >50% reduction in the monthly countable convulsive seizure frequency between 4- week Baseline period (Observational Phase) and after 12-week treatment phase using seizure diary.
  Comparing the proportion of participants with >50% reduction in the monthly countable convulsive seizure frequency between 4- week Baseline period (Observational Phase) and after 12-week treatment phase using seizure diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada